CLINICAL TRIAL: NCT06444724
Title: The Effect of Smartphone Application on the Quality of Bowel Preparation for Colonoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Uayporn Kaosombatwattana, Assistant Professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Si 422/2022
Record Dates: First submitted 2024-05-27; First posted 2024-06-05 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Colonoscopy; Bowel Preparation; Quality; Smartphone Application
Keywords: Colonoscopy; Smartphone application; Bowel preparation; Quality

STUDY DESIGN:
Intervention Model Description: Using the Line application on the smartphone to communicate with the participant
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): Patients in the control group received verbal instructions for bowel preparation before endoscopy from the endoscopy nurse, along with pamphlets containing relevant information. This instructional material encompassed details regarding a purgative regimen, instructions on its administration, dietary restrictions preceding colonoscopy, and medication adjustments necessary for some patients.
- Application group (Active Comparator): Patients in the application group will be communicated via Line applications (APP group) with guidance on preparation before colonoscopy through video media.
  Interventions: Combination Product: APP

INTERVENTIONS:
Combination Product: APP — Patients in the application group communicated via Line applications (APP group) with guidance on preparation before colonoscopy through video media.
  Other Names: Smartphone application
  Arms: Application group

SUMMARY:
The goal of this clinical trial is to learn about bowel preparation methods compared between standard techniques and enhanced education with application for elective colonoscopy. The main questions it aims to answer are:

Which bowel preparation method results in an adequate bowel preparation rate?

Participants will:

* Random to 1:1 ratio to be educated via the smartphone application (APP group) or the standard education (control group).
* Received the same purgative regimen and diet restriction.
* Endoscopist-blinded colonoscopy the participants and give score of bowel preparation scale (use Boston Bowel Preparation Scale)

DETAILED DESCRIPTION:
A prospective, endoscopist-blinded, randomized, controlled trial will conducted at the GI endoscopy center, Siriraj Hospital, Bangkok, Thailand. Patients will be divided into 2 groups in a 1:1 ratio using a computer-generated randomization method, with a block of four randomizations. Written informed consent will be obtained from all participants before their enrolment in the study.

* Patients in the control group received verbal instructions for preparation before endoscopy from the endoscopy nurse, along with pamphlets containing relevant information. This instructional material encompassed details regarding a purgative regimen, instructions on its administration, dietary restrictions preceding colonoscopy, and medication adjustments necessary for some patients.
* Patients in the application group communicated via Line applications (APP group) with guidance on preparation before colonoscopy through video media.

The registration process will entail providing basic information, including the patient's name and hospital identification number, along with the scheduled endoscopy appointment date, with strict adherence to privacy protocols. Subsequently, a trained research assistant will encourage patients to utilize the application. The video can inform the application via YouTube.

The content presented in the video corresponded identically to the verbal instructions and pamphlet provided to participants in the control group, covering topics such as the purgative regimen, dietary restrictions, and medication adjustments.

All participants will receive the same split-dose high-volume purgative regimen. Two liters of polyethylene glycol (PEG) solution regarding the composition of Colyte (hospital-based preparations) will be administered at 6-8 PM on the day before the colonoscopy, followed by 750 ml of PEG solution at 5-6 AM on the colonoscopy day.

Colonoscopies will be performed by an experienced endoscopist under intravenous sedation within 6 hours after the last preparation regimen.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 with an indication for colonoscopy
* Able to access and use Line applications on mobile phones

Exclusion Criteria:

* Patients with a history of colonic resection
* Patients with inflammatory bowel disease, polyposis syndrome, American Society of Anesthesiology (ASA) classification level 3 or higher
* Patients with a history of prior colonoscopy within 1 year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 488 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Quality bowel preparation rate | The 1 day of colonoscpy
  Quality bowel preparation will evaluated by Boston Bowel Preparation Scale score that over 6 points.

SECONDARY OUTCOMES:
Colonoscopy quality indicators : withdrawal time | During the colonoscopy
  The duration of scope withdrawal in the exception of the time used for therapeutic intervention
Colonoscopy quality indicators : polyp detection rate | During the colonoscopy
  Number of polyps detected during the scope withdrawal
Colonoscopy quality indicators : adenoma detection rate | During the colonoscopy and following the pathological result
  Number of adenoma (proof by pathology) detected during the scope withdrawal
Colonoscopy quality indicators : cecal intubation time | During the colonoscopy
  The duration of scope insertion from anus to cecum
Patient satisfaction | On the day of colonoscopy
  Evaluation of patient satisfaction with the bowel preparation protocol using the visual analog scale (Likert scale), which range from 1 (least satisfaction) to 5 (most satisfaction)
Side effects of bowel preparation | On the day of colonoscopy
  Side effects of bowel preparation will access by questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of internal medicine siriraj hospital, Mahidol university, Bangkok Noi, Bangkok, Thailand